CLINICAL TRIAL: NCT06155110
Title: Chinese People's Liberation Army General Hospital
Brief Title: A Randomized, Single-blind, Controlled Clinical Study of Cardiomyopeptidin on Improving Ischemia-reperfusion Injury in Patients With Acute ST-segment Elevation Myocardial Infarction After Primary PCI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chinese PLA General Hospital (Other)
Collaborators: Dalian Zhen-Ao Bio-Tech Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Qian geng, Clinical Professor, Chinese PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2023QG-1124
Record Dates: First submitted 2023-11-25; First posted 2023-12-04 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2023-11

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases | interventions — cardiomyopeptidin

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cardiomyopeptidin group (Experimental): The Cardiomyopeptidin group received intravenous infusion 3 mg/(kg·d) of cardiomyopeptidin during the PCI until 3 days after operation
  Interventions: Drug: cardiomyopeptidin
- The control group (No Intervention)

INTERVENTIONS:
Drug: cardiomyopeptidin — cardiomyopeptidin intervention group will accept cardiomyopeptidin (Dalian Zhenao Pharmaceutical Co., Ltd., approval number: National Drug Approval No. H20052173, specification: 20 mg/tube) 3 mg/(kg·d)；
  Arms: Cardiomyopeptidin group

SUMMARY:
This study aim to investigate the myocardium protection effect of cardiomyopeptidin in patients undergoing primary PCI for ST-elevation myocardial infarction through myocardial enhanced MRI.

DETAILED DESCRIPTION:
Investigators will enroll 160 patients with STEMI who were admitted to the Chinese PLA General Hospital between March 2022 and Marchr 2024，the investigators randomly assign eligible patients in a 1:1 ratio to either cardiomyopeptidin intervention group or control group befor primary PCI. The cardiomyopeptidin intervention group patients received intravenous infusion 3 mg/(kg·d) of cardiomyopeptidin during the PCI until 3 days after operation. Primary end point of the study was the area of infarct size measured by cardiac magnetic resonance (CMR). and secondary endpoints include slow flow/no-reflow incidence, corrected TIMI frame count (cTFC), ST-segment fall rate of ECG, cardiac enzymes and troponin, area of myocardial edema, microvascular obstruction, left ventricular ejection fraction, and composite cardiovascular events during the study period: all-cause death, cardiovascular death, unplanned hospitalization for heart failure, and revascularization. All adverse clinical events as well as study end points were monitored and adjudicated by the independent event committee.

ELIGIBILITY:
Inclusion Criteria:

* STEMI patients: typical chest pain lasting 30 min within the previous 12 h, a clear ST-segment elevation of N0.1 mV in ≥2 contiguous electrocardiographic leads, and elevated blood levels of troponin T
* patients were scheduled to undergo diagnostic cardiac angiography or percutaneous coronary interventions

Exclusion Criteria:

* had once treated by ivabradine
* history of myocardial infarction
* mechanical complications
* Unable to perform myocardial MRI
* liver and kidney failure
* malignant tumor
* unconscious
* Patients with other significant abnormal signs, laboratory tests and clinical disease are unsuitable for participation in the study accessed by clinicians.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Myocardial infarct size according to MR delayed enhancement scan | 7 days after PCI
  Two experienced MRI cardiologists analyzed the delayed enhancement image

SECONDARY OUTCOMES:
MACEs | follow up in six months
  MACEs concluding all-cause death, cardiovascular death, unplanned hospitalization for heart failure, and revascularization
myocardial edema area | 7 days after PCI
  Two experienced MRI cardiologists analyzed the delayed enhancement image
microvascular obstruction and left ventricular ejection fraction | 7 days after PCI
  Two experienced MRI cardiologists analyzed the delayed enhancement image
incidence of slow flow/no-reflow | Immediately after PCI
  Angiographic slow/no-reflow during PCI was defined as thrombolysis in myocardial infarction (TIMI) flow grade ≤ 2 during the procedure without evidence of dissection
corrected thrombolysis in myocardial infarction (TIMI) frame count (cTFC); | Immediately after PCI
  The cTFC was measured by two cardiologists, and the average value was taken. When scanning at a rate of 15 frames per second, cTFC > 20 frames per second was used as the criterion for the diagnosis of slow blood flow after primary PCI.
ST-segment fall rate of electrocardiogram (ECG) | 6 hours, 12 hours, 24 hours after myocardial infarction

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese People's Liberation Army General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Der P, Cui J, Das DK. Role of lipid rafts in ceramide and nitric oxide signaling in the ischemic and preconditioned hearts. J Mol Cell Cardiol. 2006 Feb;40(2):313-20. doi: 10.1016/j.yjmcc.2005.10.005. Epub 2005 Dec 9. PMID 16337960
- [Background] Salloum FN, Ockaili RA, Wittkamp M, Marwaha VR, Kukreja RC. Vardenafil: a novel type 5 phosphodiesterase inhibitor reduces myocardial infarct size following ischemia/reperfusion injury via opening of mitochondrial K(ATP) channels in rabbits. J Mol Cell Cardiol. 2006 Mar;40(3):405-11. doi: 10.1016/j.yjmcc.2005.10.002. Epub 2006 Feb 9. PMID 16480739
- [Background] Yang LP, Kong XP, Li RB, Zeng PL. [Recovery effect of cardiomyopeptidin fractions and fraction addition on cardiac muscle cells in rats damaged by adriamycin]. Zhongguo Zhong Yao Za Zhi. 2000 Jun;25(6):362-3. Chinese. PMID 12512426
- [Background] Yang LP, Wan HY, Kong XP, Wu Y, Teng J, Fan LL. [Preventive effect of cardiomyopeptidin on rat heart injured by ischemia-reperfusion]. Zhongguo Zhong Yao Za Zhi. 2000 Feb;25(2):105-7. Chinese. PMID 12212070
- [Background] Yang L, Chen L, Zhang G, Liu X, Chen D, Dong Y. [Effect of cardiomyopeptidin for injection on energy metabolism in isolated hearts of young rats after ischemia-reperfusion injury]. Zhong Nan Da Xue Xue Bao Yi Xue Ban. 2010 Jun;35(6):598-606. doi: 10.3969/j.issn.1672-7347.2010.06.010. Chinese. PMID 20622333
- [Background] Korosoglou G, Giusca S, Montenbruck M, Patel AR, Lapinskas T, Gotze C, Zieschang V, Al-Tabatabaee S, Pieske B, Florian A, Erley J, Katus HA, Kelle S, Steen H. Fast Strain-Encoded Cardiac Magnetic Resonance for Diagnostic Classification and Risk Stratification of Heart Failure Patients. JACC Cardiovasc Imaging. 2021 Jun;14(6):1177-1188. doi: 10.1016/j.jcmg.2020.10.024. Epub 2021 Jan 13. PMID 33454266